CLINICAL TRIAL: NCT05883124
Title: Open, Randomized, 2-period, 2-sequence, Cross-over Relative Bioavailability Study to Investigate the Pharmacokinetics and to Assess the Bioequivalence of a Rivastigmine Test Patch Formulation 9.5 mg/24 h (Twice-weekly Patch) (Luye Pharma AG, Germany) Compared to the Reference Patch Exelon® 9.5 mg/24 h (Once-daily Patch) (LTS Lohmann Therapie-Systeme AG, Germany) Applied for 11 Days
Brief Title: Rivastigmine Bioequivalence Trial With Multiple Applications of Transdermal Patches (9.5 mg/24 h)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SocraTec R&D GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1429riv22ct; 2023-000074-10 (EudraCT Number)
Record Dates: First submitted 2023-05-03; First posted 2023-05-31 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivastigmine twice-weekly 9,5 mg/24 h (Experimental): 3 consecutive applications of 1 patch (1st patch for 4 days, 2nd patch for 3 days, 3rd patch for 4 days) covering an 11-day period
  Interventions: Drug: Rivastigmine twice-weekly 9,5 mg/24 h
- Exelon® 9.5 mg/24 h (Active Comparator): 11 consecutive applications of 1 patch (each patch will be applied for 1 day) covering an 11-day period
  Interventions: Drug: Exelon® 9.5 mg/24 h

INTERVENTIONS:
Drug: Rivastigmine twice-weekly 9,5 mg/24 h — 3 consecutive applications of 1 patch (1st patch for 4 days, 2nd patch for 3 days, 3rd patch for 4 days) covering an 11-day period
  Arms: Rivastigmine twice-weekly 9,5 mg/24 h
Drug: Exelon® 9.5 mg/24 h — 11 consecutive applications of 1 patch (each patch will be applied for 1 day) covering an 11-day period
  Arms: Exelon® 9.5 mg/24 h

SUMMARY:
The present clinical trial will be conducted in order to compare the bioavailability of rivastigmine and to assess bioequivalence at steady-state of the marketed Test product Rivastigmine twice-weekly 9,5 mg/24 h transdermal patch (Manufacturer: Luye Pharma AG, Germany) and the marketed Reference product Exelon® 9.5 mg/24 h transdermal patch (Manufacturer: LTS Lohmann Therapie-Systeme AG, Germany) after multiple patch applications. Each of both treatments will last for 11 days with a washout period of at least 14 treatment-free days between the treatments.

ELIGIBILITY:
Inclusion Criteria:

1. sex: male
2. age: 18-55 years, inclusive
3. body-mass index (BMI): ≥ 18.5 kg/m² and ≤ 30.0 kg/m²
4. body weight ≥ 55 kg
5. good state of health as determined by no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination (including vital sign) and/or ECG, as determined by the investigator
6. non-smoker or ex-smoker for at least 1 month
7. written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

1. existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient (especially sick sinus syndrome or conduction defects such as sino-atrial block, atrio-ventricular block (second degree or higher)) or concomitant treatment with β-blockers
2. existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient (especially predisposition to urinary obstruction and seizures or subjects suffering from overactive bladder treated with anticholinergics)
3. existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient (especially active gastric or duodenal ulcers or predisposition to these conditions)
4. history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders, e.g. depression treated with tricyclic antidepressants, or psychosis treated with neuroleptics (cave! Metoclopramide), Parkinson's disease and predisposition to seizures
5. history of chronic obstructive or other pulmonary diseases or bronchial asthma
6. acute or history of narrow-angle glaucoma, currently treated open-angle glaucoma, or any indications from case history that there might be raised intra-ocular pressure (e.g. pressure pain, blurred vision, glaucomatous halo)
7. subjects suffering from pyloric stenosis or having difficulty in passing water owing to an impeded flow of urine (e.g. in diseases of the prostate), as well as subjects with intestinal obstruction, arrhythmia, pronounced bradycardia and severe cerebral sclerosis as well as metabolic diseases
8. known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations or previous history of application site reactions suggestive of allergic contact dermatitis with rivastigmine patch
9. history of severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
10. systolic blood pressure < 90 or > 139 mmHg
11. diastolic blood pressure < 60 or > 89 mmHg
12. heart rate < 50 bpm or > 90 bpm
13. QTc interval > 450 ms (according to Fridericia formula)
14. laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
15. ASAT > 20 % ULN, ALAT > 10 % ULN, bilirubin > 20 % ULN (except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL correspondents to of > 9 µmol/l ULN).
16. positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test and anti-HBc IgM or anti-HCV-test
17. diagnosis of COVID-19 and/or persisting disease symptoms (e.g., fever, cough) at the Investigator's discretion; current state or federal COVID-19 regulations will be considered.
18. presence or history of acute or chronic diseases especially of the skin, which could affect dermal absorption or metabolism, which may interfere with the bioavailability and /or the pharmacokinetics of the IMP or NIMP based on assessment of the investigator
19. skin abnormality (e.g. tattoo or scar) at the application site
20. acute or chronic diseases which may interfere with the pharmacokinetics of the IMP
21. history of or current drug or alcohol dependence
22. positive alcohol or drug test at screening examination
23. regular intake of alcoholic food or beverages of ≥ 24 g pure ethanol for male per day
24. subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
25. regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
26. blood donation or other blood loss of more than 400 ml within the last 6 months prior to individual enrolment of the subject
27. participation in a clinical trial with administration of any investigational medicinal product during the last 6 months prior to individual enrolment of the subject
28. simultaneous participation in another clinical trial with active ingredients
29. regular treatment with any systemically available medication (except replacement therapy, e.g. L-thyroxine)
30. subjects practising top-performance sports (more than 4 x 2 h per week)
31. close affiliation with the sponsor / the investigational site; e.g. a close relative of the investigator, dependent person (e.g. employee of or student at the investigational site), employee of the sponsor or affiliates
32. subjects suspected or known not to follow instructions
33. subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
AUC96-264 | From 96 to 264 hours after the first IMP application
  Partial area under the plasma concentration vs. time profile for the time interval 96 h 264 h
Cmax,96-264 | From 96 to 264 hours after the first IMP application
  Maximum concentration in plasma during the nominal time interval 96 h-264 h, obtained directly from measured values
CTau264 | From 96 to 264 hours after the first IMP application
  (Absolute) minimum concentration within the nominal time interval 96 h-264 h, obtained directly from measured values
Patch adhesion properties | At 96, 168 and 264 hours after the first Test patch application
  Lower one-sided 90% confidence limit for the mean of Test

SECONDARY OUTCOMES:
Adverse events | From 1st IMP application until individual discharge of a subject from the clinical trial, assessed up to approximately 2 months
  Descriptive evaluation of action taken, frequency, seriousness, intensity, relationship to the IMP/NIMP, and outcome, as well as period and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Koerner, Principal Investigator — SocraTec R&D GmbH
Locations (1):
- SocraTec R&D GmbH, Clinical Pharmacology Unit, Erfurt, Thuringia, Germany